CLINICAL TRIAL: NCT02097797
Title: Impact of Fecal transPlantAtion on MiCrobotia and hosT in Crohn's Disease
Brief Title: Impact of the Fecal Flora Transplantation on Crohn's Disease
Acronym: IMPACT-Crohn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ANRS, Emerging Infectious Diseases (Other Government); Pierre and Marie Curie University (Other); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P 121104
Record Dates: First submitted 2014-02-26; First posted 2014-03-27 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Crohn's Disease
Keywords: Inflammatory bowel disease; Crohn's disease; microbiota; fecal transplantation
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fecal Transplantation (Experimental): patients receiving the fecal transplant (fecal microbiota from a healthy donor)
  Interventions: Other: Fecal Transplantation
- Sham Transplantation (Sham Comparator): patients receiving the vehicle (Physiological serum)
  Interventions: Other: Sham Transplantation

INTERVENTIONS:
Other: Fecal Transplantation — Fecal microbiota (50-100g of stool from donor resuspended in 250-350ml of physiological serum and filtered) given by infusion in coecum during colonoscopy
  Arms: Fecal Transplantation
Other: Sham Transplantation — 250-350ml of physiological serum given by infusion in coecum during colonoscopy
  Arms: Sham Transplantation

SUMMARY:
Crohn's disease is a chronic and relapsing inflammatory bowel disease. Many data show that the intestinal flora is involved in the disease and it has been show that patients with Crohn's disease exhibit an abnormal fecal flora that might play a role in inflammation. The purpose of this study is to determine the effect of the fecal flora transplantation on Crohn's disease.

DETAILED DESCRIPTION:
Introduction : Crohn's disease (CD) is an relapsing inflammatory bowel disease relatively frequent. Its prevalence is about 1 for 700 in France, affecting predominantly young adults. Its treatment is based on immunosuppressants that might be associated with potentially severe complications such as infection and cancers. Moreover, these treatments are expensive. The gut microbiota being involved in the disease pathogenesis, it can be considered as a potential therapeutic target.

CD pathogenesis remains poorly understood but involves an inappropriate immune response toward an unbalanced gut microbiota (called dysbiosis) in predisposed hosts. The complete replacement of a dysbiotic microbiota by a "healthy" one is thus an attractive strategy. Fecal transplantation (FT) has been used with success for a long time in the context of Clostridium difficile.

Hypothesis : Fecal transplantation allow the replacement of a dysbiotic microbiota by a " healthy " one with favorable impact on CD evolution.

Primary endpoint : In CD patient with colonic or ileo-colonic involvement put in remission with corticosteroids, Evaluate if FT can modify a dysbiotic fecal microbiota to be closer of the one of a healthy donor.

Methodology

For the Receiver :

Once corticoid-induced remission will be achieved, the patient will be included and randomised to receive either FT or sham transplantation during a colonoscopy. The patient will be evaluated at week 2, 6, 10, 14, 18 and 24. At week 6, a colonoscopy will be performed.

For the Donor :

Donors will be recruited by poster advertising. When a receiver will be included, 3 donors will be contacted to attend an inclusion visit including physical examination as well as blood and stool screening for pathogen. The 3 donors will then come the day of the FT to donate their stool.

ELIGIBILITY:
Receiver

Inclusion Criteria:

* Age > 18 years and < 70 years
* Crohn's disease with colonic or ileo-colonic involvement
* Active disease at screening defined by a Harvey Bradshaw Index >4
* Clinical remission (Harvey Bradshaw Index <5) in the 3 weeks following corticosteroid onset
* Patient with health insurance
* Written consent obtained

Exclusion Criteria:

* Fistulizing disease
* Anoperineal or abdominal abscess
* Complication requiring surgical treatment
* Treatment with anti-TNFa (ongoing or stopped in the 1 month preceding randomization)
* Immunosuppressant treatment started or stopped in the 3 months preceding randomization
* Non-steroidal anti inflammatory drugs (NSAIDs) intake in the 4 weeks preceding randomization
* Antibiotics or antifungic treatment in the 4 weeks preceding colonoscopy
* Probiotics intake in the 4 weeks preceding colonoscopy
* Clostridium difficile infection in the 10 days preceding randomization
* contraindication to colonoscopy or anesthesia
* Pregnancy

Donor

Inclusion Criteria:

* Age > 20 years and < 50 years
* 27kg/m² > BMI > 17 kg/m²
* Regular bowel movement with usually one bowel movement in the morning
* Subject with health insurance
* Written consent obtained

Exclusion Criteria:

* Infection risk:

  * Known infection by human immunodeficiency virus (HIV), Human T Leukemia Virus (HTLV), Hepatitis B or C virus.
  * At risk behavior: Travel (in the preceding 3 months, excepting in Euro area, United Kingdom, Bulgaria, Poland, Romania, Croatia, Hungary, Republic Tcheque, Denmark, Norway, Sweden, Swiss, USA or Canada), at risk sexual activity (intercourse without protection with a new partner) in the preceding 6 months, blood transfusion, piercing or tattoo in the preceding 6 months residence of several years in intertropical area, abroad hospitalization more than 24 hours in the last 12 months (including patient and his immediate family).
  * Positive result at one of the screening tests for infectious disease. : HIV, HCV, HBV, HTLV, syphilis, Enteric viruses (Rotavirus, HEV, Adenovirus, Norovirus, Enterovirus, HAV, Poliovirus, Astrovirus, Aichi virus, Sapovirus), parasites in stool (Cyclospora, Isospora, Cryptosporidium, Microsporidium, Strongyloides stercoralis, Entamoeba histolitica, Giardia intestinalis, Dientamoeba fragilis), and in blood (Strongyloides stercoralis, Trichinella spiralis, Amoebiasis), pathogenic bacteria in stool (Clostridium difficile, Shigella, Campylobacter, Yersinia, Salmonella, Listeria monocytogenes, Vibrio cholerae/parahemolyticus, verotoxin-producing E. coli)
  * Anal lesions suggesting viral infection or positive test for HSV anal and/or multi-drug resistant bacteria (Enterobacteria producing extended spectrum betalactamase, Actinobacter baumanii, Vancomycin resistant enterococci and carbapenemase producing bacteria).
  * Positive test for multidrug resistant bacteria
  * If receiver is EBV negative, EBV positive donor will be excluded
  * If receiver is CMV negative, CMV positive donor will be excluded.
  * If receiver is negative for Toxoplasma gondii, positive donor for Toxoplasma gondii will be excluded
  * Known transmissible infectious disease
  * Infection (or possible infection) in the 7 days preceding screening
  * Risk factors for Creutzfeldt-Jakob disease
  * Personal history of Typhoid fever
* Gastrointestinal comorbidity

  * Personal history or first degree relative :

    * Inflammatory bowel disease
    * Coeliac disease
  * Personal history of irritable bowel syndrome, chronic constipation, chronic diarrhea
  * Personal history of gastrointestinal neoplasia or polyposis
  * First degree relative with gastrointestinal neoplasia or polyposis before 60 years old
  * Gastrointestinal infection in the 3 preceding months (defined by the occurrence of an acute diarrhea that last less than a week)
* Factors possibly affecting the composition of the microbiota:

  * Antibiotics or antifungic intake in the 3 preceding months before FT
  * Non-steroidal anti inflammatory drugs (NSAIDs) intake in the 4 weeks preceding FT
  * Specific diet (exclusion diet, vegetarian diet)
  * Pregnancy
  * Immunosuppressant intake (corticosteroids, calcineurin inhibitors, biologics, etc)
  * Anti neoplastic chemotherapy
  * Hemorrhoid disease
  * Personal history or first degree relative with inflammatory or autoimmune disease
* Other Factors :

  * Known chronic disease
  * Abnormality at initial biological check up: blood cells count, fasting, glycaemia, kidney function, liver tests, haemostasis, calprotectin
  * Long term curative therapy
  * Recent intake of food allergens related of receiver's known allergy
* between screening and FT :

  * At risk behavior (Travel, at risk sexual activity, blood transfusion, piercing tattoo, accidental blood exposure)
  * Anal lesions suggestive of viral infection or positivity for HSV in anal area
  * Infection or possible infection
  * Occurrence of gastro-intestinal symptoms
  * Medicine intake in the 48 hours preceding FT (except contraceptive)
  * In case of woman: menstruation in the 48 hours preceding FT

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-05; Primary Completion 2017-04-25 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
FT success defined by : Sorensen's index [receiver 6 weeks after FT vs donor] > Sorensen's index [receiver 6 weeks after FT vs receiver before FT]) with Sorensen's index [receiver 6 weeks after FT vs donor] ≥ 0.6. | 6 weeks after FT
  In other words, FT success is reached if the fecal microbiota of the receiver 6 weeks after FT is closer of the fecal microbiota of the donor that of the receiver before FT.
  Fecal microbiota composition will be assessed by 454 pyrosequencing (16S RNA) and microbiota comparison will be done using Sorensen's index.

SECONDARY OUTCOMES:
FT feasibility | 6 weeks after FT
  evaluate the feasibility of the FT procedure (frequency of evaluable patients in each group)
Clinical relapse rate in the 24 weeks following FT procedure | 24 weeks following FT
  Clinical relapse defined by a Crohn's disease activity index (CDAI) > 220 points, or by a CDAI between 150 and 220 with an increase >70 compared with baseline, or by the need of surgery or to start a medical treatment for CD.
Effect of FT compared to sham transplantation on CRP | 6 weeks after FT
  Effect of FT compared to sham transplantation on CRP level.
Effect of FT compared to sham transplantation on Leukocytes level | 6 weeks after FT
  Effect of FT compared to sham transplantation on: Leukocytes level
Effect of FT compared to sham transplantation on fecal calprotectin | 6 weeks after FT
  Effect of FT compared to sham transplantation on: fecal calprotectin
Effect of FT compared to sham transplantation on Crohn's Disease Endoscopic Index of Severity | 6 weeks after FT
  Effect of FT compared to sham transplantation on: Crohn's Disease Endoscopic Index of Severity
Effect of FT compared to sham transplantation on fecal microbiota composition | 6 weeks after FT
  Effect of FT compared to sham transplantation on: fecal microbiota composition
Effect of FT compared to sham transplantation on lymphocytes population in blood | 6 weeks after FT
  Effect of FT compared to sham transplantation on: lymphocytes population in blood
Effect of FT compared to sham transplantation on lymphocytes population in colon | 6 weeks after FT
  Effect of FT compared to sham transplantation on: lymphocytes population in colon.
Effect of FT compared to sham transplantation on colon transcriptomics | 6 weeks after FT
  Effect of FT compared to sham transplantation on: colon transcriptomics.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Sokol, MD, PhD, Study Director — Assistance Publique
Locations (1):
- Gastroenterology department, Saint Antoine Hospital, Paris, France

REFERENCES:
- [Derived] Sokol H, Landman C, Seksik P, Berard L, Montil M, Nion-Larmurier I, Bourrier A, Le Gall G, Lalande V, De Rougemont A, Kirchgesner J, Daguenel A, Cachanado M, Rousseau A, Drouet E, Rosenzwajg M, Hagege H, Dray X, Klatzman D, Marteau P; Saint-Antoine IBD Network; Beaugerie L, Simon T. Fecal microbiota transplantation to maintain remission in Crohn's disease: a pilot randomized controlled study. Microbiome. 2020 Feb 3;8(1):12. doi: 10.1186/s40168-020-0792-5. PMID 32014035